CLINICAL TRIAL: NCT07276698
Title: Clinical Study on Maintenance Therapy With Selinexor Combined With Azacitidine After Allogeneic Hematopoietic Stem Cell Transplantation for NK/T-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-NKT-Seli-202505
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: NK T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — selinexor; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): For patients with NK/T-cell lymphoma, maintenance therapy with selinexor combined with azacitidine was initiated 60-90 days after allogeneic hematopoietic stem cell transplantation. The specific treatment regimen was as follows:
  Selinexor 40 mg once a week; if the blood routine was intolerable (i.e., PLT ≤ 50×109/L), 20 mg once a week could be used. Azacitidine 16 mg/m2/d, days 1-5.
  A 28-day treatment cycle was adopted, and the treatment was continued for 2 years.
  Interventions: Drug: Selinexor, azacitidine

INTERVENTIONS:
Drug: Selinexor, azacitidine — For patients with NK/T-cell lymphoma, maintenance therapy with selinexor combined with azacitidine was initiated 60-90 days after allogeneic hematopoietic stem cell transplantation. The specific treatment regimen was as follows:
  Selinexor 40 mg once a week; if the blood routine was intolerable (i.e., PLT ≤ 50×109/L), 20 mg once a week could be used. Azacitidine 16 mg/m2/d, days 1-5.
  A 28-day treatment cycle was adopted, and the treatment was continued for 2 years.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation is an important treatment method for NK-T cell lymphoma, but the recurrence rate after transplantation is relatively high. Therefore, exploring efficient and low-toxicity maintenance treatment strategies after transplantation is a key challenge for improving prognosis. Previous studies have reported that selinexor and azacitidine show good anti-tumor activity in relapsed/refractory NKTCL. Thus, we conducted a single-center, single-arm, exploratory study on the efficacy and safety of selinexor combined with azacitidine as maintenance therapy after allogeneic hematopoietic stem cell transplantation for NK/T cell lymphoma, to evaluate the efficacy and safety of the combined regimen, with the aim of providing reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 18-70 years old, gender not restricted; 2. Diagnosed with NK/T-cell lymphoma (NKTCL) according to the 2022 WHO criteria; 3. Received allogeneic hematopoietic stem cell transplantation for NKTCL, with no restrictions on the type of donor; 4. Bone marrow chimerism is complete donor chimerism (T-cell chimerism > 95%); 5. ECOG: 0-1 points; 6. Blood routine must meet the following requirements: (1) ANC >= 1.0 × 10^9/L; (2) PLT >= 75 × 10^9/L; 7. The patient must be capable of understanding and willing to participate in this study, and sign the informed consent form.

Exclusion Criteria:

* 1. Those who are known to be allergic to azacitidine or selinexor; 2. Those with active acute GVHD of grade 2 or above; 3. Those with moderate or severe chronic GVHD; 4. Any unstable systemic diseases: including but not limited to unstable angina pectoris, cerebrovascular accident or transient ischemic attack (within 3 months before screening), myocardial infarction (within 3 months before screening), congestive heart failure (NYHA classification >= grade III), severe arrhythmia requiring drug treatment after pacemaker implantation, liver, kidney or metabolic diseases; patients with pulmonary hypertension. 5. Those with active uncontrolled infections: with hemodynamic instability related to infection, or new symptoms or signs of infection worsening, or new infection lesions found on imaging, persistent fever without symptoms or signs that cannot be ruled out as infection; 6. HIV-infected individuals; 7. Patients with active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral treatment; 8. History of autoimmune diseases; 9. Pregnant or lactating women; 10. Those who are currently receiving other investigational drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | two years after transplantation
over-all survival | two years after transplantation

SECONDARY OUTCOMES:
cumulative recurrence rate | one year after transplantation
cumulative recurrence rate | two years after transplantation

IPD SHARING:
Plan to Share IPD: No